CLINICAL TRIAL: NCT06203145
Title: A Clinical Study on the Whole-course Management (BCD-KPD-AutoHSCT) Scheme for Patients With Multiple Myeloma and Kidney Injury
Brief Title: A Clinical Study on the Whole-course Management (BCD-KPD-AutoHSCT) Scheme for Patients With RIMM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Yujun DONG, chief of department of hematology, Peking University First Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCD-KPD-AutoHSCT of RIMM
Record Dates: First submitted 2023-12-21; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Multiple Myeloma; Renal Injury
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; carfilzomib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BCD-KPD-AutoHSCT (Experimental): BCD-KPD-AutoHSCT/BCD-AutoHSCT
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — A reduction in serum FLCs level of more than 80% by day 14 of BCD is defined BCD-AutoHSCT group; A reduction in serum FLCs level of less than 80% by day 14 of BCD is defined BCD-KPD-AutoHSCT group.
  Other Names: Carfilzomib

SUMMARY:
Multiple myeloma (MM) is still an incurable hematological tumor, and renal involvement is the main factor of poor prognosis. The recovery of renal function can partially reverse its poor outcome. Although the 5-year survival rate of MM patients has significantly improved after entering the era of new drugs, patients with severe renal insufficiency still have a high early mortality.The purpose of this study is to investigate whether early intensive chemotherapy can reverse the proportion of renal insufficiency, is to investigate the treatment effect of RIMM patients with different renal pathological types, and is also to investigate whether autoHSCT can further partially save renal function in RIMM patients.

DETAILED DESCRIPTION:
For patients with multiple myeloma with renal impairment, the same disease stage and the same treatment regimen have different therapeutic effects. In the era of new drugs, studies have shown that early reduction of the free light chain in serum is the key to reversing renal function. The International Myeloma Working Group recommends the following drugs for the treatment of RIMM patients: 1. regimens based on proteasome inhibitors; 2. regimens based on immunomodulators. Here, we explore a clinical study on the Whole-course Management (BCD-KPD-AutoHSCT) scheme for patients with RIMM.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years or older
2. Confirmed diagnosis of symptomatic myeloma with renal impairment
3. Confirmed myeloma-associated nephropathy (e.g. light chain cast nephropathy, AL amyloidosis, MIDD etc.) on renal biopsy
4. Willingness and eligibility for autologous hematopoietic stem cell transplantation

Exclusion Criteria:

1. Pre-existing chronic kidney disease unrelated to myeloma, such as diabetic nephropathy or hypertensive nephropathy
2. Plasma cell leukemia or extramedullary plasmacytoma
3. Contraindications or prior severe allergic reactions to study medications
4. Co-existing malignancy
5. Co-existing medical conditions unsuitable for enrollment as determined by researchers, such as recent cardiovascular event, active infection etc.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-02 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
renal response rates | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided